CLINICAL TRIAL: NCT05983458
Title: Safe and Fast Discharge With Acurate Valve in Low Risk Tavi Patients
Acronym: SAFARI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Cecilia Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SAFARI
Record Dates: First submitted 2023-03-29; First posted 2023-08-09 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Stenoses, Aortic
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with severe symptomatic aortic stenosis (Other): Real-world patients with severe symptomatic aortic stenosis allocated to TAVI treatment by local heart Team will be included in the study according to the inclusion and exclusion criteria specified below.
  Interventions: Procedure: Transaortic valve replacement

INTERVENTIONS:
Procedure: Transaortic valve replacement — TAVI procedure will be performed under conscious sedation. Foley urinary catheters and jugular lines will be avoided.
  For femoral access, closure devices will be Prostar or ProGlide, which are similar and carry low rates of major vascular complications . Single femoral access and a radial access as the secondary arterial access will be used to reduce the rate of vascular complications.
  All procedures will be performed with cerebral protection using the Sentinel device. During valve implantation, commissural alignment will be checked for all patients. As a practical rule, commissural alignment will be checked in co-planar view and in cusp-overlap view.

SUMMARY:
Recent evidence from scientific literature supported the extension of TAVI procedures to lower risk populations. Despite its widespread usage, the expansion of TAVI into lower risk patient populations is still limited by complications and costs, with a large disparity between clinical trials and real-world scenarios suggesting still long hospitalizations after TAVI. This issue has got relevant implications in cost-effectiveness of the procedure, with many studies showing a more favourable cost profile associated with early discharges

DETAILED DESCRIPTION:
In most cases, prolongation of hospital stay is mainly related to electrical, renal, vascular or neurological complications. With increasing operators' experience, careful procedure planning and technology improvement, procedure-related complications are reducing, with favourable effects in terms of postprocedural length-of-stay and related costs.

This is particularly true for lower risk populations. Being surgery the gold standard for treating aortic valve disease in low-risk patients, the outcomes after TAVI in this population should meet high standards to be accepted. In particular, optimal results should not be limited to procedural success but last over time, ensuring both a long-life expectancy and a good quality of life. TAVI efficacy in this population should include the absence of residual paravalvular leaks, no need for permanent pacemakers, no cerebral embolism and the opportunity of easily re-accessing coronary arteries in the future. In particular, many questions have been raised about the difficulty of coronary re-access following use of the EvolutR/PRO valves compared to the Sapien 3 valves. Thus, valves with a larger open-celled design (ACURATE neo, Portico or JENA) are potentially more favourable for coronary access and could be considered in patients likely to require repeated re-access to coronary arteries.

Acurate Neo Valve showed good procedural results in high-risk subsets of patients. Although not tested in large-scale trials involving low risk patients, due to its unique morphology it could offer peculiar advantages, compared to other devices, including:

1. Low permanent pacemaker rates
2. Easier coronary re-access
3. Low paravalvular leak rate (novel Neo 2 technology) The aim of this study was to report on the feasibility and safety of early discharge (defined as discharge within 48 hours from the procedure) of selected low-risk patients after transfemoral TAVI with the novel Acurate Neo2 valve platform

ELIGIBILITY:
Inclusion Criteria:

1. Age >=18 and =< 83 years
2. Normal PR interval at 12-lead electrocardiogram (ECG)
3. No evidence of Right bundle branch block (RBBB) or high-degree Atrioventricular Block ( AV) blocks at 12-lead ECG
4. eGFR > 50 ml/min/1.73 m2
5. Ilio-femoral anatomy compatible with transfemoral transcatheter aortic valve implantation (TAVI)

Exclusion Criteria:

1. Inability to provide informed consent
2. Not suitable anatomy for transfemoral access
3. Need for general anaesthesia (e.g. hemodynamic instability)
4. Bicuspid aortic valve anatomy
5. Severely impaired left ventricular ejection fraction (LVEF <35%)
6. At least moderate mitral regurgitation
7. Non-cardiac illness with a life expectancy of less than 1 year
8. Currently participating in another trial before reaching first endpoint.

Ages: 18 Years to 83 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
safety and efficacy of a standardized rapid discharge protocol in low-risk patients treated with the TAVI procedure and the Acurate Neo 2 valve | 12 months
  Primary Endpoints Composite endpoints (VARC 3)
  Introduction of the composite endpoint of technical success defined at exit from procedure room with:
  freedom from mortality successful access, delivery of the device, and retrieval of the delivery system correct positioning of a single prosthetic heart valve into the proper anatomical location freedom from surgery or intervention related to the device or to a major vascular or access related, or cardiac structural complication, Expansion of device success composite endpoint at 30 days defined as: Technical Success Freedom from mortality, Freedom from surgery or intervention related to the device or to a major vascular or access-related or cardiac structural complication, Intended performance of the valve (mean gradient <20 mmHg, peak velocity <3 m/s, Doppler velocity index ≥0.25, and less than moderate aortic regurgitation) Clinical Efficacy composite endpoint now at 1 year and beyond instead of 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Nerla, MD, Principal Investigator — Maria Cecilia Hospital
Locations (1):
- Maria Cecilia Hospital, Cotignola, Ravenna, Italy

IPD SHARING:
Plan to Share IPD: No